CLINICAL TRIAL: NCT04173559
Title: Improving Perinatal Outcomes Through Activity and Sleep Tracking
Brief Title: Sleep and Tracking Effects in Pregnancy Study
Acronym: STEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of available staff
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-2434
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Complications; Pregnancy Related; Weight Gain; Weight Change Trajectory; High Risk Pregnancy; Stress, Emotional
MeSH Terms: conditions — Pregnancy Complications; Weight Gain; Body-Weight Trajectory; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Women randomized to this group will receive no guidance regarding exercise / activity / sleep during pregnancy.
- Activity Intervention (Experimental): Women randomized to this group will receive detailed information and reminders about physical activity and sleep in pregnancy. .
  Interventions: Behavioral: Activity Intervention

INTERVENTIONS:
Behavioral: Activity Intervention — After 1 week of baseline activity is obtained, participants will be contacted with personalized activity goals that are 10% higher than their previous weeks' activity levels. They will also receive feedback regarding sleep if they are not averaging at least 6 hours per night or if they are waking more than twice per night. Participants will also receive weekly text reminders and encouraging feedback, and will receive additional counseling in person at regularly scheduled prenatal visits until delivery.
  Arms: Activity Intervention

SUMMARY:
Purpose: The investigators hypothesize that a simple, personalized, smartphone-based activity intervention using a wrist-based activity tracker will help high risk pregnant women reduce their stress during pregnancy.

Participants: Pregnant women enrolled in prenatal care at the University of North Carolina who have a documented moderate or high level of perceived stress ( ≥ 14) and are at high risk for adverse pregnancy outcomes due to body mass index of ≥ 30 kg/m2 or history of gestational hypertension, preeclampsia, intrauterine growth restriction, or preterm birth <37 weeks' in a prior pregnancy.

Procedures: Women meeting inclusion criteria will be recruited through the University of North Carolina prenatal care clinics. They will be contacted for possible participation at regularly scheduled prenatal visits and/or ultrasound. They may also be contacted for possible participation by remote methods (e.g., Telehealth). Women who are enrolled will complete validated dietary, stress, sleep, and body image questionnaires. Enrolled women will then be randomized to receive standard obstetrical care or enhanced counseling. All participants will receive a wrist-based activity tracker. Maternal blood sample for biochemical markers of stress and gene expression will be obtained at the initial visit; a followup blood sample will be obtained later in pregnancy, and a small portion of the placenta saved at delivery. Maternal and neonatal outcomes will be compared between groups.

DETAILED DESCRIPTION:
During pregnancy, women regularly interact with healthcare professionals, an often untapped resource and opportune time to minimize stress and optimize weight gain, nutrition, and activity, positively impacting outcomes and lifelong health. The overarching hypothesis of this study is that a simple, personalized, smartphone-based activity intervention using a wrist-based activity tracker will help high risk pregnant women increase their activity level during pregnancy, reduce stress, and optimize gestational weight gain and biometric parameters. Importantly, the investigators propose that women can be engaged in care via a simple, personalized text-message based intervention.

Women will be enrolled early in pregnancy and followed prospectively. All women will receive a wrist-based activity tracker. Some women (those randomized to receive individualized counseling) will receive weekly text messages based on their activity and sleep in the prior week. Other women will not receive any specific instructions regarding activity level. The investigators will follow their outcomes prospectively. Biologic samples (including blood, urine, vaginal swabs, placental tissue) will be collected at enrollment and at delivery.

ELIGIBILITY:
Inclusion Criteria:

* At high risk for adverse pregnancy outcomes, due to either body mass index ≥ 30 kg/m^2, or a prior history of preeclampsia, intrauterine growth restriction or preterm birth prior to 37 weeks' gestation in a previous pregnancy and a perceived stress score of >/= 14 (10-question scale)
* Gestational age of 8.0 to 19.9 weeks' gestation using American College of Obstetricians and Gynecologists dating criteria (combination of ultrasound and menstrual dating, as available)
* Current singleton viable intrauterine pregnancy. Spontaneous reduction of twin to singleton gestation is allowable provided it occurred prior to 14 weeks' gestation.
* No structural abnormalities or aneuploidy
* Ability to communicate in and provide consent in English
* Maternal age 18 to 51 years of age
* Owns smartphone compatible with wrist-based activity tracker (over 200 devices supported)

Exclusion Criteria:

* Women pregnant with multifetal gestations
* Women who have a medical condition where a modest increase in low-impact activity is contraindicated (at the discretion of the woman's treating physician)
* Planned delivery prior to 36 weeks' of gestation
* Unwilling to wear wrist-based activity tracker for at least 6 out of 7 days per week

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05-14 (Estimated); Study Completion 2025-05-14 (Estimated)

PRIMARY OUTCOMES:
Reduction in Perceived Maternal Stress | through delivery, an average of 7 months per participant
  Perceived stress score will be calculated using a validated 10-question stress scale; score = 14 indicates moderate stress
Proportion of women with adverse perinatal outcomes | outcome will be ascertained at delivery
  The investigators will define adverse pregnancy outcomes as a composite of preterm birth <37 weeks, intrauterine growth restriction, preeclampsia, and placental abruption; outcomes will be compared between randomization groups.

SECONDARY OUTCOMES:
Number of activity goals met by personalized activity level group | through delivery, an average of 7 months per participant
  Proportion of weekly activity goals that were successfully met by women randomized to personalized activity group
Mean Daily steps | through delivery, an average of 7 months per participant
  Mean number of daily steps; amount will be compared between randomization groups.
Median Daily steps | through delivery, an average of 7 months per participant
  median number of daily steps; amount will be compared between randomization groups.
Mean 'Moderate' or greater physical activity | through delivery, an average of 7 months per participant
  Mean number of weekly minutes of 'moderate' or 'intense' physical activity as registered by the wrist-based activity monitor; amount will be compared between randomization groups.
Median 'Moderate' or greater physical activity | through delivery, an average of 7 months per participant
  median number of weekly minutes of 'moderate' or 'intense' physical activity as registered by the wrist-based activity monitor; amount will be compared between randomization groups.
Mean Nightly sleep minutes | through delivery, an average of 7 months per participant
  Mean number of sleep minutes per night; amount will be compared between randomization groups.
Median Nightly sleep minutes | through delivery, an average of 7 months per participant
  median number of sleep minutes per night; amount will be compared between randomization groups.
Median resting heart rate parameters | through delivery, an average of 7 months per participant
  The change in the median resting heart rate level and nadir of the resting heart rate (in beats per minute), between enrollment and delivery ; amount will be compared between randomization groups.
Mean Resting heart rate parameters | through delivery, an average of 7 months per participant
  The change in the mean resting heart rate level and nadir of the resting heart rate (in beats per minute), between enrollment and delivery ; amount will be compared between randomization groups.
Median Body composition change during study - total body water | through reassessment of body composition at 16 weeks after randomization, an average of 4 months per participant.
  The change in median total body water measurements between enrollment and re-assessment at 8 and 16 weeks (as applicable, if still pregnant) after enrollment will be compared between randomization groups.
Mean Body composition change during study - total body water | through reassessment of body composition at 16 weeks after randomization, an average of 4 months per participant.
  The change in mean total body water measurements between enrollment and re-assessment at 8 and 16 weeks (as applicable, if still pregnant) after enrollment will be compared between randomization groups.
Median Body composition change during study - percent body fat | through reassessment of body composition at 16 weeks after randomization, an average of 4 months per participant.
  The change in median percent body fat measurements between enrollment and re-assessment at 8 and 16 weeks (as applicable, if still pregnant) after enrollment will be compared between randomization groups.
Mean Body composition change during study - percent body fat | through reassessment of body composition at 16 weeks after randomization, an average of 4 months per participant.
  The change in mean percent body fat measurements between enrollment and re-assessment at 8 and 16 weeks (as applicable, if still pregnant) after enrollment will be compared between randomization groups.
Gestational weight gain | through delivery, an average of 7 months per participant
  The amount of weight gained by each participant during pregnancy, in pounds. outcomes will be compared between randomization groups.
Gestational weight gain, per week after study enrollment | through delivery, an average of 7 months per participant
  The amount of weight gained per week by each participant, in pounds, between study enrollment and delivery. outcomes will be compared between randomization groups.
Proportion of women with gestational diabetes mellitus | through delivery, an average of 7 months per participant.
  The diagnosis of gestational diabetes mellitus during pregnancy, using standard criteria as set forth by American College of Obstetricians and Gynecologists. outcomes will be compared between randomization groups.
Proportion of women with hypertensive complications of pregnancy | through 6 weeks' postpartum, an average of 7 months per participant
  The diagnosis of gestational hypertension, preeclampsia, or eclampsia, using standard American College of Obstetricians and Gynecologists diagnostic criteria. outcomes will be compared between randomization groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy A Manuck, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol
Time Frame: 12 to 36 months after initial publication
Access Criteria: Access will be given provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Olson CM, Strawderman MS, Reed RG. Efficacy of an intervention to prevent excessive gestational weight gain. Am J Obstet Gynecol. 2004 Aug;191(2):530-6. doi: 10.1016/j.ajog.2004.01.027. PMID 15343232
- [Background] Muktabhant B, Lumbiganon P, Ngamjarus C, Dowswell T. Interventions for preventing excessive weight gain during pregnancy. Cochrane Database Syst Rev. 2012 Apr 18;4(4):CD007145. doi: 10.1002/14651858.CD007145.pub2. PMID 22513947
- [Background] Muktabhant B, Lawrie TA, Lumbiganon P, Laopaiboon M. Diet or exercise, or both, for preventing excessive weight gain in pregnancy. Cochrane Database Syst Rev. 2015 Jun 15;2015(6):CD007145. doi: 10.1002/14651858.CD007145.pub3. PMID 26068707
- [Background] Wolf HT, Owe KM, Juhl M, Hegaard HK. Leisure time physical activity and the risk of pre-eclampsia: a systematic review. Matern Child Health J. 2014 May;18(4):899-910. doi: 10.1007/s10995-013-1316-8. PMID 23836014
- [Background] Sorensen TK, Williams MA, Lee IM, Dashow EE, Thompson ML, Luthy DA. Recreational physical activity during pregnancy and risk of preeclampsia. Hypertension. 2003 Jun;41(6):1273-80. doi: 10.1161/01.HYP.0000072270.82815.91. Epub 2003 Apr 28. PMID 12719446